CLINICAL TRIAL: NCT06298903
Title: The Effect of a Hip Activation Home Exercise Program (HEP) Compared to a Hip Activation + Single Leg Balance HEP on the Forward Step-Down Test in Healthy Females
Brief Title: Impact of Hip Activation Compared to Hip Plus Balance Training on the Forward-Step-Down Test
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Louisiana State University Health Sciences Center Shreveport (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00002565
Record Dates: First submitted 2024-01-19; First posted 2024-03-07 (Actual); Last update posted 2024-12-13 (Actual); Status verified 2024-12

CONDITIONS: Control of Frontal Plane Biomechanics; Patellofemoral Pain Syndrome
MeSH Terms: conditions — Patellofemoral Pain Syndrome

STUDY DESIGN:
Who Masked: Investigator
Masking Description: The investigator who will analyze the data will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hip activation (Active Comparator): Participants will perform a hip muscle activation program 2 days per week for 8 weeks. The HEP consists of 5 exercises that target the gluteal muscles.
  Interventions: Other: Hip Activation
- Hip activation + Single leg balance (Experimental): Participants will perform a hip muscle activation program as in the active comparator group, plus a single leg balance training HEP 2 days per week for 8 weeks. The hip HEP consists of 5 exercises that target the gluteal muscles. The single leg balance HEP consists of a variety of eyes open and eyes closed single leg balance exercises.
  Interventions: Other: Hip activation + Single leg balance

INTERVENTIONS:
Other: Hip Activation — Sidelying hip abduction, side plank with hip abduction, clamshell (hip abduction + external rotation), side plan with clamshell, and quadruped fire hydrant exercises will be performed for 1 minute isometric holds, 2 times per week for 8 weeks.
  Arms: Hip activation
Other: Hip activation + Single leg balance — Hip activation HEP: Sidelying hip abduction, side plank with hip abduction, clamshell (hip abduction + external rotation), side plan with clamshell, and quadruped fire hydrant exercises will be performed for 1 minute isometric holds, 2 times per week for 8 weeks.
  Single leg balance: variety of single leg balance exercises with different upper extremity and lower extremity positions to provide different balance stimuli. Weeks are alternated performing these exercises with eyes open and eyes closed.
  Arms: Hip activation + Single leg balance

SUMMARY:
The purpose of this research is to determine the impact of a hip activation home exercise program (HEP) compared to a hip activation + single leg balance HEP on performance of the Forward-Step-Down Test (FSDT) in healthy females. Participants will be assigned to the control (hip activation HEP only) or experimental (hip activation + single leg balance HEP). Following the pre-test data collection, participants will complete their HEP for 8 weeks. They will return to the lab for post-test measurements.

ELIGIBILITY:
Inclusion Criteria:

* first or second year students at the institutions's School of Allied Health Professions
* healthy
* female

Exclusion Criteria:

* participating in another research study
* current knee pain or pathology on the dominant leg
* known diagnosis of vestibular impairment
* known pregnancy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2024-01-12 (Actual); Primary Completion 2024-03-25 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Forward-Step-Down Test | pre-intervention (baseline), post-intervention (8 weeks)
  a step-down task that is performed off a 20 cm box. Five repetitions are performed to give one score (minimum score 0, maximum score 6). A higher score is worse.

SECONDARY OUTCOMES:
surface electromyography (sEMG) peak | pre-intervention (baseline), post-intervention (8 weeks)
  The peak sEMG will be collected from the dominant side's gluteus maximum and gluteus medius muscles. The sEMG will be collected during both the FSDT and unipedal stance test
surface electromyography (sEMG) mean | pre-intervention (baseline), post-intervention (8 weeks)
  The mean sEMG will be collected from the dominant side's gluteus maximum and gluteus medius muscles. The sEMG will be collected during both the FSDT and unipedal stance test
Unipedal Stance Test (UPST) | pre-intervention (baseline), post-intervention (8 weeks)
  The time a participant can stand on one leg will be collected for eyes open and eyes closed conditions.
Dose-Response | post-intervention (8 weeks)
  The dose-response for outcome 1, 2, and 3 will be calculated, using participant's self-reported exercise compliance as the dose.

CONTACTS AND LOCATIONS:
Overall Officials: Erin McCallister, DPT, Principal Investigator — LSUHSC-Shreveport
Locations (1):
- LSUHSC-Shreveport, Shreveport, Louisiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cannon J, Weithman BA, Powers CM. Activation training facilitates gluteus maximus recruitment during weight-bearing strengthening exercises. J Electromyogr Kinesiol. 2022 Apr;63:102643. doi: 10.1016/j.jelekin.2022.102643. Epub 2022 Feb 9. PMID 35189569
- [Background] Rinaldi VG, Prill R, Jahnke S, Zaffagnini S, Becker R. The influence of gluteal muscle strength deficits on dynamic knee valgus: a scoping review. J Exp Orthop. 2022 Aug 17;9(1):81. doi: 10.1186/s40634-022-00513-8. PMID 35976534
- [Background] Wilczynski B, Zorena K, Slezak D. Dynamic Knee Valgus in Single-Leg Movement Tasks. Potentially Modifiable Factors and Exercise Training Options. A Literature Review. Int J Environ Res Public Health. 2020 Nov 6;17(21):8208. doi: 10.3390/ijerph17218208. PMID 33172101
- [Background] Khayambashi K, Mohammadkhani Z, Ghaznavi K, Lyle MA, Powers CM. The effects of isolated hip abductor and external rotator muscle strengthening on pain, health status, and hip strength in females with patellofemoral pain: a randomized controlled trial. J Orthop Sports Phys Ther. 2012 Jan;42(1):22-9. doi: 10.2519/jospt.2012.3704. Epub 2011 Oct 25. PMID 22027216
- [Background] Khayambashi K, Fallah A, Movahedi A, Bagwell J, Powers C. Posterolateral hip muscle strengthening versus quadriceps strengthening for patellofemoral pain: a comparative control trial. Arch Phys Med Rehabil. 2014 May;95(5):900-7. doi: 10.1016/j.apmr.2013.12.022. Epub 2014 Jan 16. PMID 24440362
- [Background] Hott A, Liavaag S, Juel NG, Brox JI. Study protocol: a randomised controlled trial comparing the long term effects of isolated hip strengthening, quadriceps-based training and free physical activity for patellofemoral pain syndrome (anterior knee pain). BMC Musculoskelet Disord. 2015 Feb 25;16:40. doi: 10.1186/s12891-015-0493-6. PMID 25879452
- [Background] Hewett TE, Myer GD, Ford KR. Decrease in neuromuscular control about the knee with maturation in female athletes. J Bone Joint Surg Am. 2004 Aug;86(8):1601-8. doi: 10.2106/00004623-200408000-00001. PMID 15292405
- [Background] Lee SP, Powers CM. Individuals with diminished hip abductor muscle strength exhibit altered ankle biomechanics and neuromuscular activation during unipedal balance tasks. Gait Posture. 2014 Mar;39(3):933-8. doi: 10.1016/j.gaitpost.2013.12.004. Epub 2013 Dec 12. PMID 24373699
- [Background] Hatton AL, Kemp JL, Brauer SG, Clark RA, Crossley KM. Impairment of dynamic single-leg balance performance in individuals with hip chondropathy. Arthritis Care Res (Hoboken). 2014 May;66(5):709-16. doi: 10.1002/acr.22193. PMID 24115764
- [Background] Alfuth M, Gomoll M. Electromyographic analysis of balance exercises in single-leg stance using different instability modalities of the forefoot and rearfoot. Phys Ther Sport. 2018 May;31:75-82. doi: 10.1016/j.ptsp.2018.01.002. Epub 2018 Mar 21. PMID 29573984
- [Background] Anguish B, Sandrey MA. Two 4-Week Balance-Training Programs for Chronic Ankle Instability. J Athl Train. 2018 Jul;53(7):662-671. doi: 10.4085/1062-6050-555-16. PMID 30192681
- [Background] Rothermel S, Hale S, Hertel J, Denegar C. Effect of active foot positioning on the outcome of a balance training program. Physical Therapy in Sport. 2004. 5:2 (98-103). https://doi.org/10.1016/j.ptsp.2004.02.002.
- [Background] McCallister E, Flowers DW. Can the Forward-Step-Down Test Be Used Reliably in the Clinical Setting to Assess Movement Changes Resulting from Maximal Exertion? A Pilot Study. The Internet Journal of Allied Health Sciences and Practice. 2020 Jan 01;18(4), Article 7. doi: 10.46743/1540-580X/2020.1931
- [Background] Hopper AJ, Haff EE, Joyce C, Lloyd RS, Haff GG. Neuromuscular Training Improves Lower Extremity Biomechanics Associated with Knee Injury during Landing in 11-13 Year Old Female Netball Athletes: A Randomized Control Study. Front Physiol. 2017 Nov 7;8:883. doi: 10.3389/fphys.2017.00883. eCollection 2017. PMID 29163219
- [Background] McGovern RP, Martin RL, Christoforetti JJ, Kivlan BR. EVIDENCE-BASED PROCEDURES FOR PERFORMING THE SINGLE LEG SQUAT AND STEP-DOWN TESTS IN EVALUATION OF NON-ARTHRITIC HIP PAIN: A LITERATURE REVIEW. Int J Sports Phys Ther. 2018 Jun;13(3):526-536. PMID 30038839
- [Background] Fisher BE, Southam AC, Kuo YL, Lee YY, Powers CM. Evidence of altered corticomotor excitability following targeted activation of gluteus maximus training in healthy individuals. Neuroreport. 2016 Apr 13;27(6):415-21. doi: 10.1097/WNR.0000000000000556. PMID 26981714
- [Background] Loudon JK, Wiesner D, Goist-Foley HL, Asjes C, Loudon KL. Intrarater Reliability of Functional Performance Tests for Subjects With Patellofemoral Pain Syndrome. J Athl Train. 2002 Sep;37(3):256-261. PMID 12937582
- [Background] Springer BA, Marin R, Cyhan T, Roberts H, Gill NW. Normative values for the unipedal stance test with eyes open and closed. J Geriatr Phys Ther. 2007;30(1):8-15. doi: 10.1519/00139143-200704000-00003. PMID 19839175
- [Background] Flowers DW, Brewer W, Mitchell K, Ellison J, Frilot C. The Effect of Core Stabilization Training on Improving Gait and Self-Perceived Function in Patients with Knee Osteoarthritis: A Single-Arm Clinical Trial. Pathophysiology. 2022 Sep 1;29(3):495-506. doi: 10.3390/pathophysiology29030040. PMID 36136067
- [Background] Clark L, Dean A, Mitchell A, & Torgerson DJ. Envelope use and reporting in randomised controlled trials: a guide for researchers. Research Methods in Medicine & Health Sciences. 2021;2(1):2-11. doi:10.1177/2632084320957204
- [Background] van Melick N, Meddeler BM, Hoogeboom TJ, Nijhuis-van der Sanden MWG, van Cingel REH. How to determine leg dominance: The agreement between self-reported and observed performance in healthy adults. PLoS One. 2017 Dec 29;12(12):e0189876. doi: 10.1371/journal.pone.0189876. eCollection 2017. PMID 29287067
- [Background] Konrad P. The ABC of EMG: A Practical Introduction to Kinesiological Electromyography.
- [Background] Distefano LJ, Blackburn JT, Marshall SW, Padua DA. Gluteal muscle activation during common therapeutic exercises. J Orthop Sports Phys Ther. 2009 Jul;39(7):532-40. doi: 10.2519/jospt.2009.2796. PMID 19574661
- [Background] Selkowitz DM, Beneck GJ, Powers CM. Comparison of Electromyographic Activity of the Superior and Inferior Portions of the Gluteus Maximus Muscle During Common Therapeutic Exercises. J Orthop Sports Phys Ther. 2016 Sep;46(9):794-9. doi: 10.2519/jospt.2016.6493. Epub 2016 Aug 5. PMID 27494053
- [Background] Harput G, Ulusoy B, Akmese R, Ergun N. Comparison of muscle activation levels and knee valgus between individuals with medial patellofemoral ligament reconstruction and healthy individuals during fatiguing step down task. Clin Biomech (Bristol). 2020 Aug;78:105067. doi: 10.1016/j.clinbiomech.2020.105067. Epub 2020 Jun 6. PMID 32535475
- [Background] Selkowitz DM, Beneck GJ, Powers CM. Which exercises target the gluteal muscles while minimizing activation of the tensor fascia lata? Electromyographic assessment using fine-wire electrodes. J Orthop Sports Phys Ther. 2013 Feb;43(2):54-64. doi: 10.2519/jospt.2013.4116. Epub 2012 Nov 16. PMID 23160432
- [Background] Chan MK, Chow KW, Lai AY, Mak NK, Sze JC, Tsang SM. The effects of therapeutic hip exercise with abdominal core activation on recruitment of the hip muscles. BMC Musculoskelet Disord. 2017 Jul 21;18(1):313. doi: 10.1186/s12891-017-1674-2. PMID 28732494
- [Background] Henry KD, Rosemond C, Eckert LB. Effect of number of home exercises on compliance and performance in adults over 65 years of age. Phys Ther. 1999 Mar;79(3):270-7. PMID 10078770
- [Background] Eckard T, Lopez J, Kaus A, Aden J. Home exercise program compliance of service members in the deployed environment: an observational cohort study. Mil Med. 2015 Feb;180(2):186-91. doi: 10.7205/MILMED-D-14-00306. PMID 25643386